CLINICAL TRIAL: NCT06246071
Title: A Phase Ia/Ib, Multicenter, Open-label Study of TYK-00540, Administered Orally in Adult Patients With Locally Advanced/Metastatic Solid Tumors
Brief Title: A Study of TYK-00540 in Adult Patients With Solid Tumors
Acronym: ASOTIAPWST
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TYKM5807102
Record Dates: First submitted 2024-01-18; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-12

CONDITIONS: Locally Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TYK-00540 (Experimental): Escalation stage: Multiple doses of TYK-00540 tablets as monotherapy for oral administration to find the maximum tolerated dose. The administration frequency will be twice daily (BID), every 28 days as a cycle.
  Expansion stage: an optimal dose of TYK-00540 tablets for cohort expansion. The administration frequency will be twice daily (BID), every 28 days as a cycle.
  Interventions: Drug: TYK-00540

INTERVENTIONS:
Drug: TYK-00540 — TYK-00540 PO, BID

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of TYK-00540, with dose-escalation stage and dose-expansion stage.

DETAILED DESCRIPTION:
To evaluate dose limiting toxicities (DLT) and determine the maximum tolerated dose (MTD) in subjects with locally advanced or metastatic solid tumors.

To investigate the pharmacokinetic profile of TYK-00540 and its metabolites after single then multiple doses of TYK-00540 administered orally once daily. To assess preliminary effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. In the Single-agent escalation phase, subjects should fulfill the following criterion at Screening: Histologically or cytologically confirmed locally advanced/metastatic solid tumors that do not have, failed or intolerated standard of care (SOC).In the single-agent expansion phase, subjects should fulfill the following criteria at Screening: Cohort 1: Histologically or cytologically confirmed platinum-resistant HGSOC (Platinum-resistant: responds at first to treatment with drugs that contain platinum, but then comes back within 6 months period; only female subjects will be enrolled). Cohort 2: Histologically or cytologically confirmed locally advanced/metastatic TNBC who have received two lines of standard of care (SOC) regimens, including:

   1. Any prior treatment can be considered as one of the SOC regimens if executed on patients with the receptor status of triple-negative no matter the previous pathological type;
   2. For patients whose treatment have been changed due to intolerability to toxicity, the intolerable regimens can be included as one of the prior standards of care regimens;
   3. For neoadjuvant and/or adjuvant chemotherapy, if relapse or disease progression to locally advanced or metastatic disease occurs during treatment or within 12 months after discontinuation of treatment (at least 2 cycles have been completed), it will be considered as one of the SOC regimens;
   4. For patients with documented germline BRCA1/BRCA2 mutations, if they have been treated with an approved PARP inhibitor, then the PARP inhibitor can be considered as one of the 2 lines of prior SOC regimens required.

   In the combination-agent escalation and combination expansion phase (Cohort 3), subjects should fulfill the following criteria at Screening: ER+/HER2-breast cancer with who have relapsed or progressed after treatment with CDK4/6 inhibitors (no prior treatment of fulvestrant or other SERDs, SERCA; no contraindications to the use of fulvestrant; for locally advanced or metastatic disease stages, the number of chemotherapy lines≤ 1). Note: Histologically-confirmed breast carcinoma expressing positive ER (≥1% tumor cells expressing ER as positive on IHC staining, recommended by ASCO/CAP Guideline Update 2020. For the purposes of the expansion study, only ER+ IHC staining ≥10% will be considered ER+ in this cohort. Negative HER2 is defined as IHC 0 or 1+, or IHC 2+ but confirmed by the negative ISH, recommended by ASCO/CAP Guideline 2018.
3. Subjects in the escalation phase should have measurable or evaluable lesions at baseline; Measurable lesions required in the expansion phase (RECIST 1.1).
4. ECOG performance status is 0 to 1 and there is no deterioration in the 2 weeks prior to the first dose.
5. Life expectancy of at least 3 months.
6. Adequate organ functions, defined as: ALT or AST ≤ 2.5×the upper limit of normal (ULN) or ≤ 5 ×ULN with documented liver involvement (such as liver metastasis or a primary biliary tumor) and Total bilirubin ≤ 1.5 ×ULN (subjects with Gilbert's Disease may be enrolled with Sponsor approval); Absolute neutrophil count (ANC) ≥ 1.5×109/L, Platelet count ≥ 80 ×109/L and Hemoglobin (Hb) ≥ 9 mg/dL, not requiring growth factor and transfusion support for at least 14 days prior to screening; Adequate renal function, creatinine clearance ≥ 60 mL/min (According to the Cockcroft and Gault formula). Coagulation function: International normalized ratio (INR) ≤ 1.5 ×ULN and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN. Left ventricular ejection fraction (LVEF) ≥50%.
7. Willing and able to provide written informed consent approved by institutional review board (IRB) or independent ethics committee (IEC).
8. Willingness of men and women of reproductive potential to observe conventional and effective birth control for the duration of treatment and 6 months following the last dose of study treatment; this may include barrier methods such as condom or diaphragm with spermicidal gel.

Exclusion Criteria:

1. Known allergy to any excipients of TYK-00540 tablets (for combination-agent escalation phase and combination expansion phase, known contraindications to fulvestrant should also be considered).
2. Subjects with prior therapy of: Systemic anti-tumor treatment such as standard chemotherapy, macromolecular targeted drugs and immunological drug therapy within 28 days prior to the first dose; reception of endocrine therapy, small molecule targeted drugs and oral fluorouracil within 14 days before the first dose; reception of nitrosoureas and mitomycin within 6 weeks prior to the first dose Major surgery (except minor surgeries such as appendicitis and tumor biopsy) within 4 weeks prior to the planned start of TYK-00540. Subjects who have taken proton pump inhibitors (PPIs) within 7 days prior to the first dose of TYK-00540, or require continuation of therapy during the study. Subjects who were receiving and need to continue treatment with medications known to prolong the QTc interval or potentially cause Torsade de pointe ventricular tachycardia during the treatment. Participation in other clinical trials (excluding non-interventional drug clinical trials) within 28 days prior to the first dose; Prior allogeneic bone marrow transplantation.
3. Subjects with other malignancies or a history of other malignant tumors, except for cured basal cell carcinoma of the skin or squamous cell carcinoma, carcinoma in situ of the cervix, papillary thyroid cancer, carcinoma in situ of the breast duct, or other malignant tumors that have survived for more than 5 years.
4. Any unresolved toxicities from prior therapy greater than NCI CTCAE Grade 1 at the time of starting study treatment with the exception of Grade 2 alopecia and prior platinum-therapy related neuropathy.
5. Patients with primary central nervous system (CNS) tumors or CNS metastases that have failed local therapy. Patients who are asymptomatic or clinically stable and do not require steroids and other treatments for CNS metastases ≥ 28 days and are radiographically stable during the screening period may be enrolled.
6. The subject has symptoms of spinal cord compression due to the tumor.
7. Uncontrollable or poorly controlled effusion of chest, abdomen, pelvis, or pericardium.
8. Any baseline 12-lead ECG abnormalities which may impair the safety of subjects (such as baseline QTc interval ≥ 470 msec, complete left bundle branch block (LBBB), acute or unspecified myocardial infarction, active myocardial ischemic ST-T segment changes with clinical significance, second- or third-degree atrioventricular (AV) block, or severe bradycardia or tachycardia).
9. Have had any of the following in the past 6 months: myocardial infarction, long QT syndrome, torsades de pointes, arrhythmias (double-bundle branch block, such as right bundle branch block (RBBB) with left anterior or posterior branch block, third-degree atrioventricular block) , unstable angina, coronary/peripheral artery bypass grafting, symptomatic chronic heart failure (CHF), Grade III or IV cardiac function as defined by the New York Heart Association, cerebrovascular accident, transient cerebral ischemia, symptomatic pulmonary embolism, and/or other clinically significant thromboembolic disease episodes. NCI CTCAE ≥ Grade 2 persistent arrhythmia, any grade of atrial fibrillation (asymptomatic uncomplicated atrial fibrillation was required to be of ≥Grade 2). Enrollment of patients who have an implanted cardiac rhythm device/pacemaker with QTcF > 470 msec needs to be discussed by the investigators and sponsor.
10. Subjects with any other disease or medical condition that is unstable or could affect their safety or study compliance, any serious or uncontrolled systemic disease, including uncontrolled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg). Uncontrolled diabetes, active bleeding, ocular lesions, and other serious mental, neurological, cardiovascular or respiratory system diseases.
11. Known active infections, including human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV) infection, except for asymptomatic chronic HBV or HCV carriers. Active HBV, HCV, or HIV infections are defined as:

    1. Hepatitis B surface antigen (HBsAg) positive and HBV-DNA ≥ 2000 cps/mL or 500 IU/mL; HBsAg-negative, anti-HBc-positive patients are at high risk of HBV reactivation who require suppressive antiviral therapy prior to initiation of cancer therapy;
    2. Anti-HCV antibody positive and HCV-RNA > upper normal limit defined by sites;
    3. Anti-HIV antibody positive with uncontrolled opportunistic infections; anti-HIV antibody positive with CD4+ count< 350 cells/uL that requires HIV therapy prior to the cancer treatment; other conditions allowing concurrent ART but the therapy not tolerated and that the toxicities confused with investigational drug toxicities.
12. History of positively diagnosed interstitial lung disease or interstitial pneumonia (ILD), drug-induced ILD, or radiation pneumonitis requiring hormone therapy, or any evidence of active ILD (e.g., acute onset or progressive pneumonitis/pulmonary fibrosis at baseline), or the pulmonary symptoms which are not suitable for enrollment in the investigator's judgment or the high-risk factors which may cause interstitial lung disease and are not suitable for enrollment.
13. Clinically significant gastrointestinal abnormalities at screening that may affect the intake, transport or absorption of drugs (such as dysphagia, uncontrollable nausea and vomiting, active gastric ulcer, ulcerative colitis, Crohn's disease, chronic diarrhea, intestinal obstruction, gastric diseases requiring long-term administration of PPIs without a cure, etc.).
14. Clinically significant hypercoagulability.
15. Pregnant and lactating women.
16. Subjects who, in the opinion of the investigator, would not be suitable for participation in this study (e.g., not in line with the treatment of the subject's best benefit, subject compliance, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Within 31 days of the first dose
  Numbers of participants experiencing AEs which are defined as DLTs classfied by CTCAE
Recommended dose for combination-agent escalation and single-agent expansion (RDE) | 1 year
  To determine the recommended dose for combination-agent escalation and single-agent expansion agent expansion.
Adverse events (AEs) | From Baseline up to 28 days after the end of the treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Objective response rate (ORR) | At least 24 weeks
  ORR is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) assessment in accordance to Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

SECONDARY OUTCOMES:
The time to the peak concentration (Tmax) | 0 hours (h) (within 30 min before dosing), 0.25 h, 0.5 h , 1 h , 2 h , 3 h, 4 h, 8 h , 12 h, 24 h after dosing
  Tmax is defined as the time of maximum concentration of the drug in blood observed after a drug dose administration.
Maximum plasma concentration (Cmax) | 0 hours (h) (within 30 min before dosing), 0.25 h, 0.5 h , 1 h , 2 h , 3 h, 4 h, 8 h , 12 h, 24 h after dosing
  Cmax is the maximum (or peak) plasma concentration that the drug achieves in blood after the drug has been administered.
Minimum plasma concentration (Cmin) | 0 hours (h) (within 30 min before dosing), 0.25 h, 0.5 h , 1 h , 2 h , 3 h, 4 h, 8 h , 12 h, 24 h after dosing
  Cmin is the minimum plasma concentration that the drug achieves in blood after the drug has been administered.
Area under the plasma concentration time | 0 hours (h) (within 30 min before dosing), 0.25 h, 0.5 h , 1 h , 2 h , 3 h, 4 h, 8 h , 12 h, 24 h after dosing
  AUC0-inf defined as the area under the plasma concentration-time curve from time 0 extrapolated to Infinite time.
Disease Control Rate (DCR) | At least 24 weeks
  DCR is defined as the proportion of patients with a best overall response of complete response (CR) , partial response (PR) or Stable disease (SD) ≥6 weeks during the study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Hospital, Hefei, China

IPD SHARING:
Plan to Share IPD: No